CLINICAL TRIAL: NCT04546958
Title: Clinical Implication of Nutritional Counseling and Whey Protein Supplements in Patients on Peritoneal Dialysis with Hypoalbuminemia
Brief Title: Nutritional Interventions in Peritoneal Dialysis Patients with Hypoalbuminemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wan-Chuan Tsai, Principal Investigator, Assistant Professor, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FEMH-IRB-109116-F
Record Dates: First submitted 2020-09-06; First posted 2020-09-14 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: End Stage Renal Disease on Dialysis
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: A randomized, active-controlled trial with cross-over design
Who Masked: Outcomes Assessor
Masking Description: Laboratory technicians who assess the study outcomes will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutritional counseling arm (Active Comparator): Nutritional counseling, targeting daily protein intake 1.2 g/kg Dietitian will provide one-to-one dietary education, 30 minutes duration, on a monthly basis
  Interventions: Other: Nutritional counseling
- Nutritional counseling plus whey protein supplements arm (Experimental): Nutritional counseling plus whey protein supplements, targeting daily protein intake 1.5 g/kg In addition to receiving nutritional counseling, participants are instructed to take an additional whey protein supplement at the dose of ~0.3 g/kg protein intake.
  Interventions: Dietary Supplement: Whey protein supplements; Other: Nutritional counseling

INTERVENTIONS:
Dietary Supplement: Whey protein supplements — Nutritional counseling and whey protein supplements for 3 months
  Arms: Nutritional counseling plus whey protein supplements arm
Other: Nutritional counseling — Nutritional counseling by dietitians for 3 months

SUMMARY:
Inadequate dietary protein intake is well-known cause of hypoalbuminemia in dialysis population. Protein loss into dialysate and increased catabolic state due to uremic milieu or inflammation worsened hypoalbuminemia, hence high protein diet is recommended in patients on peritoneal dialysis (PD). The recommendations from K/DOQI clinical practice guidelines for the amount of daily protein intake is based on expert opinion and the optimal daily protein intake in PD patients is not known. The investigators hypothesize that higher dietary protein intake has a greater beneficial effect on nutritional status in hypoalbuminemic PD patients. In particular, 1.5 g/kg protein intake provides a better beneficial effect than 1.2 g/kg protein intake.

DETAILED DESCRIPTION:
Hypoalbuminemia is common and is strongly associated with an increased risk for mortality in patients with end-stage kidney disease (ESKD). Inadequate dietary protein intake is well-known cause of hypoalbuminemia in dialysis population. Protein loss into dialysate and increased catabolic state due to uremic milieu or inflammation worsened hypoalbuminemia, hence high protein diet is recommended in PD patients. Although there is an increased daily calorie intake from absorption of dialysate glucose concentration, hypoalbuminemia ensues in a substantial number of PD patients. There is concern that a disproportionately increasing calorie intake from dialysate glucose with no change in dietary protein intake causes weight gain which in turn worsens sarcopenic obesity in PD patients. Achieving adequate dietary protein intake should be the priority in the management of hypoalbuminemia. It is feasible for PD patients to increase dietary protein intake through protein supplements. Among nutritional supplements, whey protein has several positive effects on carbohydrate metabolism, muscle building, immune function, and human health in various areas of disease, supported by well-performed studies. There are limited data available regarding the effects of nutritional counseling and whey protein supplements on the nutritional, body compositional status and immune function of PD patients with hypoalbuminemia. The recommendations from K/DOQI clinical practice guidelines for the amount of daily protein intake is based on expert opinion and the optimal daily protein intake in PD patients is not known.

The aims of the study are to investigate the optimal dietary protein intake and to examine the effects of whey protein supplement on the change of nutritional, body composition and immune function in PD patients with hypoalbuminemia. Specifically, the investigators will compare the effect of nutritional counseling (1.2 g/kg protein intake) with that of nutritional counseling and whey protein supplement (1.5 g/kg protein intake) regarding the changes of nutritional, body composition parameters and immune function in PD patients. This is a quality improvement program to cope with the fact that the proportion of hypoalbuminemic PD patients sometimes does not meet the requirements set by Joint Commission of Taiwan, and to improve the nutritional status of PD patients in a feasible way of daily clinical practice.

The investigators are going to conduct a randomized, controlled trial with cross-over design. Subjects with ESKD undergoing maintenance PD for more than three months, adequate dialysis, and hypoalbuminemia will be recruited. Those with non-dietary cause of hypoalbuminemia including untreated fluid overload, uncorrected metabolic acidosis, having active infection or inflammation, hospitalization within the past 4 weeks, having gastrointestinal bleeding, those who cannot cooperate with the dietary record, those who have poor adherence to whey protein consumption, history of psychiatric disorders and having mental retardation will be excluded. Participants will receive nutritional counseling with whey protein supplement or nutritional counseling alone for 3-month period, separated by 3-month washout period. The study outcome measures are difference in change-from-baseline nutritional, body composition parameters and immune function between the two study periods.

ELIGIBILITY:
Inclusion Criteria:

1. Aged greater than or equal to 20 years
2. Having end-stage kidney disease and having undergone maintenance PD for more than three months
3. Having adequate dialysis (weekly Kt/V greater than or equal to 1.7)
4. Serum albumin levels lower than 4.0 g/dL, measured by bromocresol green assay

Exclusion Criteria:

1. Untreated fluid overload
2. Uncorrected metabolic acidosis
3. Having active infection or inflammation
4. Hospitalization within the past 4 weeks
5. Having gastrointestinal bleeding
6. those who cannot cooperate with the dietary record
7. those who have poor adherence to whey protein consumption
8. History of psychiatric disorders
9. Having mental retardation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Concentrations of albumin (g/dL) | 3 months
  Difference in change-from-baseline albumin (g/dL) between two intervention arms

SECONDARY OUTCOMES:
Concentrations of pre-albumin (g/dL) | 3 months
  Difference in change-from-baseline pre-albumin (g/dL) between two intervention arms
Concentrations of C-reactive protein (mg/dL) | 3 months
  Difference in change-from-baseline C-reactive protein (mg/dL) between two intervention arms
Concentrations of phosphate (mg/dL) | 3 months
  Difference in change-from-baseline phosphate (mg/dL) between two intervention arms
Concentrations of blood urea nitrogen (mg/dL) | 3 months
  Difference in change-from-baseline blood urea nitrogen (mg/dL) between two intervention arms
Concentrations of free indoxyl sulfate (mg/L) | 3 months
  Difference in change-from-baseline free indoxyl sulfate (mg/L) between two intervention arms
Concentrations of free p-cresol sulfate (mg/L) | 3 months
  Difference in change-from-baseline free p-cresol sulfate (mg/L) between two intervention arms
Absolute number (per μl blood) of CD4+ (cluster of differentiation 4) T cells | 3 months
  Difference in change-from-baseline absolute number (per μl blood) of CD4+ T cells between two intervention arms
Absolute number (per μl blood) of CD8+ (cluster of differentiation 8) T cells | 3 months
  Difference in change-from-baseline absolute number (per μl blood) of CD8+ T cells between two intervention arms
Absolute number (per μl blood) of monocytes | 3 months
  Difference in change-from-baseline absolute number (per μl blood) of monocytes between two intervention arms
Percentage (%) of CD4+ (cluster of differentiation 4) T cells | 3 months
  Difference in change-from-baseline percentage (%) of CD4+ T cells between two intervention arms
Percentage (%) of CD8+ (cluster of differentiation 8) T cells | 3 months
  Difference in change-from-baseline percentage (%) of CD8+ T cells between two intervention arms
Percentage (%) of monocytes | 3 months
  Difference in change-from-baseline percentage (%) of monocytes between two intervention arms
Lean tissue mass (kg) | 3 months
  Difference in change-from-baseline lean tissue mass (kg) between two intervention arms
Fat tissue mass (kg) | 3 months
  Difference in change-from-baseline fat tissue index (kg) between two intervention arms
Lean tissue index (kg/m2) | 3 months
  Difference in change-from-baseline lean tissue index (kg/m2) between two intervention arms
Fat tissue index (kg/m2) | 3 months
  Difference in change-from-baseline fat tissue index (kg/m2) between two intervention arms
Percentage (%) of body fat mass | 3 months
  Difference in change-from-baseline percentage (%) of body fat mass between two intervention arms
Percentage (%) of excess body fat | 3 months
  Difference in change-from-baseline percentage (%) of excess body fat between two intervention arms. Excess body fat is defined as fat percentage > 25 % for men or > 35 % for women
Percentage (%) of obesity | 3 months
  Difference in change-from-baseline percentage (%) of obesity between two intervention arms. Obesity is defined as body mass index > 24.

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Chuan Tsai, M.D., Ph.D., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Individual-level deidentified participant data will be made available by the corresponding author of the paper upon request by email. The data will be available for 3 years after formal publication.
Supporting Information: Study Protocol
Time Frame: The data will become available after completing the study for 1 year and for 3 years after formal publication.
Access Criteria: Data will be made available by the corresponding author of the paper upon request by email.